CLINICAL TRIAL: NCT07270731
Title: Investigation of Safety, Tolerability, Pharmacokinetic and Pharmacodynamics of Single Administrations of NNC9733-0001 in Healthy Participants and in Participants With Type 2 Diabetes
Brief Title: A Research Study of a New Medicine, NNC9733-0001, in Healthy Participants and Participants With Type 2 Diabetes
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NN9733-8133; U1111-1314-8868 (Other: World Health Organization (WHO)); 2024-519382-22 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteer; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC9733-0001 (Experimental): Participants will be administered a single dose of NNC9733-0001 in a dose escalated manner.
  Interventions: Drug: NNC9733-0001
- Placebo (Experimental): Participants will be administered a single dose of matching NNC9733-0001 placebo in a dose escalated manner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC9733-0001 — Administered a single dose of NNC9733-0001.
  Arms: NNC9733-0001
Drug: Placebo — Administered a single dose of matching NNC9733-0001 placebo.
  Arms: Placebo

SUMMARY:
This study is testing a new medicine that might help treat people with type 2 diabetes. The study is conducted to see if the new medicine can lower high sugar levels in the blood. The purpose of the study is to see if the new study medicine is safe and how well is tolerated by the body. There will be two groups of partici-pants in this study: healthy participants and participants with type 2 diabetes. Participant will either get study medicine (NNC9733-0001) or placebo (a treatment that has no active medicine in it). Which treatment the participant gets is decided by chance. Which dose (strength) the participant get is determined by when participant enter the study. Participant will get one dose which will be injected into the area around abdomen (belly) by the medical staff. The number of injections (up to 4 injections) will depend on the group the participant is assigned to. Larger doses require multiple injections. The study will last for about 40 weeks (10 months).

ELIGIBILITY:
Inclusion Criteria:

All participants

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine eligibility for the study.
* Male, or female of nonchildbearing potential

Healthy participants

* Age 18-45 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2) (both inclusive) at screening.
* Glycosylated haemoglobin (HbA1c) less than or equal to (≤) 6.4 percent (%) (47 millimoles per mole (mmol/mol)) at screening.
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, Electrocardiography (ECG), and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Participants with T2DM

* Age 18-64 years (both inclusive) at the time of signing the informed consent.
* BMI between 20.0 and 34.9 kg/m^2 (both inclusive) at screening.
* HbA1c 6.5-8.5% (47.5-69.4 mmol/mol) at screening.
* Diagnosed with type 2 diabetes mellitus (T2DM) greater than or equal to (≥) 180 days before screening.
* Stable daily dose(s) of metformin within 90 days before screening.

Exclusion Criteria:

* Screening alanine transaminase (ALT) values greater than (>) upper limit of normal (ULN) +10 per-cent (%), AST values >ULN +20%, or total bilirubin >ULN.
* Renal impairment, defined as estimated glomerular filtration rate (eGFR) less than (<) 60.0 millilitre per minute per 1.73-meter square (mL/min/1.73m^2), at screening.
* Clinical evidence of Chronic Kidney Disease (CKD) and/or urinary albumin:creatinine ratio (UACR) >30 milligram per gram (mg/g).
* Presence or history of cardiovascular disease, including stable and unstable angina pectoris, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias, or clinically significant conduction disorders.

Healthy participants

* Any disorder, which in the investigator's opinion, might jeopardise participants' safety or compliance with the protocol.
* Supine blood pressure at screening outside the range of 90-139 millimetres of mercury (mmHg) for systolic or 50-89 mmHg for diastolic.

Participants with T2DM - Any disorder, except for mild conditions under stable treatment associated with T2DM, which in the investigator's opinion might jeopardise participant safety or compliance with the protocol.

• Supine blood pressure at screening outside the range of 90-159 mmHg for systolic or 50-99 mmHg for diastolic. This exclusion criterion also pertains to those participants who are receiving antihypertensive treatment.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From dosing (day 1) until end of study (EOS) visit (week 36)
  Measured as number of events
Number of hypoglycaemic events | From dosing (day 1) until end of study (EOS) visit (week 36)
  Measured as number of events

SECONDARY OUTCOMES:
AUC0-last: The area under the NNC9733-0001 plasma concentration-time curve from time zero to last measurable concentration after a single dose | From dosing (day 1) to 48 hours after dosing
  Measured in hours × nanogram/millilitre (ng/mL)
Cmax: The maximum concentration of NNC9733-0001 in plasma | From dosing (day 1) to 48 hours after dosing
  Measured in nanogram/millilitre (ng/mL)
tmax: The time from dose administration to maximum plasma concentration of NNC9733-0001 | From dosing (day 1) to 48 hours after dosing
  Measured in hours
t1/2: Terminal half-life for NNC9733-0001 after a single dose | From dosing (day 1) to 48 hours after dosing
  Measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com